CLINICAL TRIAL: NCT07379320
Title: Validity and Reliability of the Multidimensional Scale of Perceived Social Support in Individuals With Lower Extremity Amputation
Brief Title: Psychometric Evaluation of the Multidimensional Scale of Perceived Social Support in Lower Extremity Amputation
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Erbahceci, Professor, Hacettepe University
Other Study IDs: FTREK25-161
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lower Limb Amputation
Keywords: Lower limb amputation; Perceived social support; Psychometric validation; Reliability; Validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Limb Amputation Cohort: This cohort includes adults aged 18 years and older with lower extremity amputation who are recruited during routine clinical follow-up visits. Participants will complete questionnaires assessing perceived social support and related psychosocial outcomes.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational study. No therapeutic or behavioral intervention is administered. Participants only complete questionnaire-based assessments.

SUMMARY:
The purpose of this study is to examine the validity and reliability of the Multidimensional Scale of Perceived Social Support in individuals with lower extremity amputation. Social support plays an important role in psychological well-being, social participation, and adaptation after amputation. However, there is limited evidence regarding whether this scale accurately and consistently measures perceived social support in individuals with lower limb amputation.

Participants aged 18 years and older with lower extremity amputation will be invited to complete several questionnaires, including the Multidimensional Scale of Perceived Social Support. Some participants will complete the social support questionnaire a second time within a short period to evaluate the consistency of the results. The findings of this study are expected to contribute to the accurate assessment of perceived social support in individuals with lower limb amputation and to support future clinical and research applications.

DETAILED DESCRIPTION:
This methodological study aims to evaluate the validity and reliability of the Turkish version of the Multidimensional Scale of Perceived Social Support in individuals with lower extremity amputation. Perceived social support is a key psychosocial factor influencing psychological adjustment, social participation, and quality of life following amputation. Although the Multidimensional Scale of Perceived Social Support has been validated in various populations, its psychometric properties have not been sufficiently examined in individuals with lower limb amputation.

Individuals aged 18 years and older with lower extremity amputation will be recruited from routine clinical follow-up visits. Participants will complete a sociodemographic data form and standardized questionnaires assessing perceived social support, psychosocial adjustment, participation, and health-related quality of life. To assess test-retest reliability, the Multidimensional Scale of Perceived Social Support will be re-administered to a subgroup of participants within a 3 to 7-day interval.

Reliability will be evaluated using internal consistency and test-retest reliability analyses. Construct validity will be examined through correlations between perceived social support scores and related psychosocial and health measures. The results of this study will provide evidence regarding the psychometric adequacy of the Multidimensional Scale of Perceived Social Support for use in individuals with lower extremity amputation and will support its application in both clinical practice and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and older.
* Individuals with unilateral or bilateral lower extremity amputation.
* Ability to read and understand Turkish.
* Ability to provide informed consent and complete self-reported questionnaires.

Exclusion Criteria:

* Presence of severe cognitive impairment or neurological disorders that may affect comprehension of the questionnaires.
* Presence of acute psychiatric conditions that may interfere with participation.
* Presence of additional medical conditions that significantly limit communication or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years and older with lower extremity amputation who are attending routine clinical follow-up visits. Participants are individuals who are able to communicate in Turkish and who consent to participate in questionnaire-based assessments related to perceived social support and psychosocial outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of the Multidimensional Scale of Perceived Social Support | Baseline and 3-7 days
  The validity and reliability of the Multidimensional Scale of Perceived Social Support will be evaluated using internal consistency, test-retest reliability, and construct validity analyses in individuals with lower extremity amputation.

SECONDARY OUTCOMES:
Psychosocial adjustment assessed by the Trinity Amputation and Prosthesis Experience Scales | Baseline
  Psychosocial adjustment, activity restriction, and prosthesis satisfaction will be assessed using the Trinity Amputation and Prosthesis Experience Scales in individuals with lower extremity amputation.
Participation level assessed by the Reintegration to Normal Living Index | Baseline
  Participation in daily and social life will be assessed using the Reintegration to Normal Living Index.
Health-related quality of life assessed by the Nottingham Health Profile | Baseline
  Health-related quality of life will be assessed using the Nottingham Health Profile.

IPD SHARING:
Plan to Share IPD: No